CLINICAL TRIAL: NCT05606120
Title: A Post-market Study Evaluating Clinical and Radiographic Early Outcomes of Hip Arthroplasty With CL TRAUMA Cemented Femoral Stem
Brief Title: H-35 CL TRAUMA Cemented Femoral Stem
Status: Completed | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-35
Record Dates: First submitted 2022-10-19; First posted 2022-11-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty; Replacement; Hip
Keywords: Hip replacement; Cemented stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CL TRAUMA implanted patients: Patients who underwent hip arthroplasty with CL TRAUMA cemented femoral stem from 2017 to 2023.
  Interventions: Device: CL TRAUMA femoral stem

INTERVENTIONS:
Device: CL TRAUMA femoral stem — Hip arthroplasty according to the instruction for use.

SUMMARY:
Study design: monocentric, retrospective, observational and post-market clinical study.

Purpose: To demonstrate the safety and performance of CL TRAUMA femoral stem. The eligible study population is represented by the entire population that underwent a hip replacement with CL TRAUMA femoral stem from 2017 to 2023 at Azienda Ospedaliera di Padova (IT) in accordance with the indication for use of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Age > 18 years old;
3. All patients must give written informed consent approved by the study site's Institutional Review Board (IRB)/Ethical Committee (EC);
4. Adult patients in whom a decision has already been made to perform a partial or total hip arthroplasty with CL TRAUMA femoral stem as per indication for use. The decision to implant CL TRAUMA must be taken prior to, and independently from the decision to enroll the patient. This decision should be made in accordance with routine clinical practice at the study site concerned;
5. Patients suffering from: non-inflammatory degenerative joint disease including osteoarthritis, avascular necrosis and dysplasia; or suffering from rheumatoid arthritis; or patients requiring treatment of femoral head and neck fractures;
6. Patients able to comply with the protocol.

Exclusion Criteria:

1. Adult patients with any CL TRAUMA femoral stem contraindication for use as reported in the current local Instruction for use;
2. Patients with active or any suspected infection (on the affected hip or systemic);
3. Patients suffering from acute or chronic osteomyelitis;
4. Patients with confirmed nerve or muscle lesion compromising hip joint function;
5. Patients with vascular or nerve diseases affecting the concerned limb;
6. Patients with poor bone stock (such as osteoporosis or extended previous revision surgery) compromising the stability of the implant;
7. Patients with metabolic disorders which may impair fixation and stability of the implant;
8. Any concomitant disease and dependence that might affect the implanted prosthesis;
9. Patients with known incompatibility or allergy to the product materials, and/or metal hypersensitivity to implant materials;
10. Patients currently participating in any other surgical intervention studies or pain management studies;
11. Female patients who are pregnant, nursing or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible study population is represented by the entire population that underwent a hip replacement with CL TRAUMA femoral stem from 2017 to 2023.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is based upon Harris Hip score evaluation. | Performed only at survival follow-up (up to 7 years).
  The primary endpoint is based upon patients' clinical recovery at the Survival Follow-up visit measured as Harris Hip Score greater than 80.
  The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery, and it is intended to evaluate various hip disabilities and methods of treatment in an adult population. It is a clinical outcome measurement administered by a qualified health care professional, such as a physician or a physical therapist. There are ten items covering four domains. The domains are: pain, function, absence of deformity, and range of motion.
  The maximum score is 100 points. Results can be interpreted with the following:
  * < 60 = failed result;
  * 60-69 = poor result;
  * 70-79 = fair;
  * 80-90 = good
  * 90-100 = excellent.

SECONDARY OUTCOMES:
Radiographic implant evaluation and stability assessment at different routinely post-operative timepoints. | Performed at discharge, 1 month follow-up, 2 years follow-up and at survival follow-up (up to 7 years).
  Imaging will be collected to evaluate the radiographic performance of the device, which will contribute to the overall efficacy evaluation of the CL TRAUMA femoral stem.
  All X-rays performed during the clinical study fall within standard clinical practice.
  Radiological assessment was carried out postoperatively at discharge, at 1 month and 24 months after the surgery. It included standard views, such as antero-posterior (AP) of the pelvis and lateral (LAT) of the affected hip.
Survivorship of the implant (Kaplan-Meier estimate) after surgery at survival follow-up. | Performed only at survival follow-up (up to 7 years).
  The Kaplan-Meier estimate for implant revision will be calculated and shown graphically. The time from the initial operation to the revision date will be described in person-years, and the Poisson incidence rate and associated 95% CI (confidence interval) will be provided.
Safety assessment | From surgery to survival follow-up (up to 7 years).
  Incidence, type and severity of all the Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Padova, Italy